CLINICAL TRIAL: NCT03997929
Title: Prospective Evaluation of 1.3-ß-D-glucan in the Peritoneal Fluid for the Diagnosis of Fungal Peritonitis in Critically Ill Patients
Brief Title: Peritoneal 1.3-ß-D-glucan for the Diagnosis of Intra-abdominal Candidiasis in Critically Ill Patients (pBDG2)
Acronym: pBDG2
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI074
Record Dates: First submitted 2019-05-09; First posted 2019-06-25 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-02

CONDITIONS: Intra Abdominal Infections; Candidiasis, Invasive; Peritoneal Candidiasis; Critically Ill
MeSH Terms: conditions — Intraabdominal Infections; Candidiasis, Invasive; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CASE (intra abdominal candidiasis): Critically ill patients with a confirmed diagnosis of intra abdominal candidiasis (IAC) Definition of IAC : sterilely collected peritoneal fluid cultures that are positive for Candida spp. as determined by the signs and symptoms consistent with an active infection
  Interventions: Diagnostic Test: 1.3 BETA D GLUCAN
- CONTROL (bacterial intra abdominal infection): Critically ill patients with a non candida intra abdominal infection (bacterial peritonitis)
  Interventions: Diagnostic Test: 1.3 BETA D GLUCAN

INTERVENTIONS:
Diagnostic Test: 1.3 BETA D GLUCAN — dosage of 1.3 BETA D GLUCAN in the peritoneal fluid obtained during surgery with the β-glucan test (Fujifilm Wako Chemicals, Osaka, Japan)

SUMMARY:
New rapid diagnostic strategies are warranted in intra-abdominal candidiasis (IAC). A previous retrospective study showed that one measure, the day of the surgery, of peritoneal 1.3-Beta-D-Glucan ≤ 310pg/ml could rule out an IAC. This strategy was independent of the patient underlying conditions and Candida risk factors. This study aimed to confirm these results with a multicenter prospective study

ELIGIBILITY:
Inclusion Criteria:

* critically ill adult (> 18 yrs old) admitted to ICU for intra-abdominal infection requiring surgery and possible intra abdominal candidiasis

Exclusion Criteria:

* declinate to participate,
* expected death within the first 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of 200 patients. Among them, identification of : 50 Cases (confirmed intra abdominal candidiasis) and 50 controls (intra abdominal infection without candida).
  If more than 50 cases, random selection. Identification of control by matching (with confounding factors of the 1.3 BDG test). If more than 50 controls after matching, random selection.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Measure of 1.3 BDG in the peritoneal exudate of patient with intra-abdominal candidiasis | 1 DAY
  Value of 1.3 BDG in the peritoneal exudate in patient with intra-abdominal candidiasis in comparison with non intra-abdominal candidiasis

SECONDARY OUTCOMES:
Measure of 1.3 BDG in the serum of patient with intra-abdominal candidiasis | DAY 1 and DAY 3
  Coefficient of correlation between peritoneal and serum 1.3 BDG in patient with and without intra-abdominal candidiasis

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel NOVY, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (4):
- France (4):
  - CHR Mercy, Metz, Lorraine
  - PILI-FLOURY Sebastien, Besançon
  - BOUHEMAD Belaid, Dijon
  - POTTECHER Julien, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Available from inclusion to end of participation of the included patient
Access Criteria: Only access to IPD of patient of the own participating ICU Access by code

REFERENCES:
- [Background] Novy, E.; Laithier, F.-X.; Riviere, J.; Remen, T.; Losser, M.-R.; Guerci, P.; Machouart, M. Protocol for the pBDG2 Study: Prospective Evaluation of 1.3-β-D-Glucan in the Peritoneal Fluid for the Diagnosis of Intra-Abdominal Candidiasis in Critically Ill Patients. Microbiol. Res. 2021, 12, 196-203. https://doi.org/10.3390/microbiolres12010015
- [Result] Novy E, Laithier FX, Machouart MC, Albuisson E, Guerci P, Losser MR. Determination of 1,3-beta-D-glucan in the peritoneal fluid for the diagnosis of intra-abdominal candidiasis in critically ill patients: a pilot study. Minerva Anestesiol. 2018 Dec;84(12):1369-1376. doi: 10.23736/S0375-9393.18.12619-8. Epub 2018 Jul 9. PMID 29991219